CLINICAL TRIAL: NCT01501708
Title: Phase II Study of Caspofungin Based Combined Anti-fungal Therapy for Patients With Proven or Probable Invasive Fungal Infection After Allogeneic Stem Cell Transplantation From HLA-matched Unrelated or HLA-mismatched Related Donors
Brief Title: Caspofungin Based Combined Anti-fungal Therapy for Proven or Probable Invasive Fungal Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, M.D., Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-2011-71
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia; Transplantation, Hematopoietic Stem Cell
Keywords: caspofungin; IFI; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia | interventions — Caspofungin; Voriconazole; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caspofugin based combination therapy (Experimental): Caspofugin based combination therapy:
  Patients will recieve caspofungin with voriconazole or amphotericin B
  Interventions: Drug: Caspofugin based combination therapy

INTERVENTIONS:
Drug: Caspofugin based combination therapy — Caspofungin: 70 mg on the ﬁrst day of therapy, followed by 50 mg q.d.
  * All patients received azoles as prophylaxis (fluconazole as prophylaxis and itraconazole or voriconazole as secondary prophylaxis), combination with liposomal amphotericin B at a dosage 3mg/kg q.d will be given.
  * In case of renal function damage, combination with voriconazole 6mg/kg followed by 4 mg/kg b.i.d. will be given.
  Other Names: caspofungin + voriconazole or amphotericin B

SUMMARY:
In this prospective phase II observational study, we plan to assess the efficacy and tolerability of caspofungin based combined anti-fungal therapy for proven or probable IFI in a group of patients received allo-HSCT transplantation with high risk of IFI: HLA matched unrelated donor or mismatched donor conditioning with ATG containing regimen or present III-IV aGVHD or extensive GVHD undergoing high-dose steroid treatment.

DETAILED DESCRIPTION:
Patients will recieve caspofungin with either voriconazole or amphotericin B as combination therapy for fungal infection

ELIGIBILITY:
Inclusion Criteria:

* adult patient undergoing allogeneic hematopoietic stem cell transplantation
* age 18-55 years
* with inform consent
* no contraindication for allogeneic transplantation: active infection, allergy to FLu/Bu/CTX, liver and renal function damage
* HLA mismatched related (3~5/6) or unrelated donors (at least 8/10)
* proven or probable IFI

Exclusion Criteria:

* age less than 18 years or over 56 years
* HLA mismatched related donor
* liver function/renal function damage (over 2 X upper normal range)
* with mental disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Favorable response rate | 12 weeks

SECONDARY OUTCOMES:
Overall survival | 12 weeks, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ling Wang, M.D., Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No